CLINICAL TRIAL: NCT00086801
Title: Phase II Trial of Doxorubicin, Vinblastine, and Gemcitabine (AVG) Chemotherapy for Non-Bulky Stage I and II Hodgkin's Lymphoma
Brief Title: Combination Chemotherapy in Treating Patients With Newly Diagnosed Stage I or Stage II Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-50203; U10CA031946 (NIH); CALGB-50203; CDR0000370870 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Lymphoma
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Doxorubicin; Gemcitabine; Vinblastine; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- doxorubicin + vinblastine + gemcitabine (Experimental): Patients receive doxorubicin IV over 3-5 minutes, vinblastine IV over 3-5 minutes, and gemcitabine IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Patients undergo fludeoxyglucose F 18 positron-emission tomography (PET) scanning and CT scan before treatment and after courses 2 and 6 of therapy to assess response. Patients with a positive PET scan after completion of study therapy may undergo biopsy. A PET scan is performed 3 months later if biopsy is negative or biopsy is unable to be performed.
  Patients are followed every 3 months for 1 year, every 4 months for 2 years, every 6 months for 2 years, and then annually for 5 years.
  Interventions: Drug: doxorubicin hydrochloride; Drug: gemcitabine hydrochloride; Drug: vinblastine; Procedure: fludeoxyglucose F 18 positron-emission tomography (PET) scan; Procedure: CT scan

INTERVENTIONS:
Drug: doxorubicin hydrochloride — given IV
Drug: gemcitabine hydrochloride — given IV
Drug: vinblastine — given IV
Procedure: fludeoxyglucose F 18 positron-emission tomography (PET) scan
Procedure: CT scan

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin, vinblastine, and gemcitabine, work in different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: This phase II trial is studying how well combination chemotherapy works in treating patients with newly diagnosed stage I or stage II Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the complete response rate in patients with newly diagnosed stage IA, IB, IIA, or IIB non-bulky Hodgkin's lymphoma treated with doxorubicin, vinblastine, and gemcitabine.

Secondary

* Determine the event-free survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Determine whether fludeoxyglucose F 18 positron-emission tomography scanning is useful in predicting clinical relapse and determining the presence of residual disease in these patients after treatment with this regimen.

OUTLINE: This is a multicenter study.

Patients receive doxorubicin IV over 3-5 minutes, vinblastine IV over 3-5 minutes, and gemcitabine IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo fludeoxyglucose F 18 positron-emission tomography (PET) scanning and CT scan before treatment and after courses 2 and 6 of therapy to assess response. Patients with a positive PET scan after completion of study therapy may undergo biopsy. A PET scan is performed 3 months later if biopsy is negative or biopsy is unable to be performed.

Patients are followed every 3 months for 1 year, every 4 months for 2 years, every 6 months for 2 years, and then annually for 5 years.

ELIGIBILITY:
1. Documentation of Disease:

   1.1 Histologically documented Hodgkin lymphoma subclassified according to the WHO modification of the Rye Classification and staged according to the modified Ann Arbor Staging Classification system. Patients must have clinical stage IA, IB, IIA or IIB. Patients with "E" extensions will be eligible if all other criteria have been met. Nodular lymphocyte predominant Hodgkin lymphoma is excluded.
   * Core biopsies are acceptable if they contain adequate tissue for primary diagnosis and immunophenotyping. Fine needle aspirate (FNA) cytologies and bone marrow biopsies as the sole means of diagnosis are not acceptable.
   * Note: Failure to submit pathology slides within 60 days of patient registration will result in patient being declared ineligible.

   1.2 Patients may not have a mediastinal mass > 0.33 maximum intrathoracic diameter on standing postero-anterior chest x-ray or peripheral or retroperitoneal adenopathy > 10 cm in its largest diameter.

   1.3 Bone marrow biopsy is required for pretreatment evaluation. Bilateral biopsies are preferred but not required.
2. No prior treatment (chemotherapy or radiation therapy) for Hodgkin lymphoma.
3. Measurable disease must be present either on physical examination or imaging studies. Any tumor mass measurable in two dimensions and > 2 cm is acceptable (or 1.5 cm if 0.5 cm slices are used as in spiral CT scans). Lesions that are considered intrinsically non-measurable include the following:

   * bone lesions
   * leptomeningeal disease
   * ascites
   * pleural/pericardial effusion
   * inflammatory breast disease
   * lymphangitis cutis/pulmonis
   * abdominal masses that are not confirmed and followed by imaging techniques
   * cystic lesions
   * lesions that are situated in a previously irradiated area
4. Age ≥ 16 years
5. Performance status 0-2
6. LVEF by ECHO or MUGA within institutional normal limits
7. DLCO ≥ 60% with no symptomatic pulmonary disease
8. No known HIV infection. Patients with a history of intravenous drug abuse or any behavior associated with an increased risk of HIV infection should be tested for exposure to the HIV virus. Patients who test positive or who are known to be infected are not eligible due to an increased risk of infection with this chemotherapy regimen. An HIV test is not required for entry on this protocol, but is required if the patient is perceived to be at risk.
9. Non-pregnant and non-lactating. Due to the teratogenic potential of the agents used in this study, pregnant or nursing women may not be enrolled. Women and men of reproductive potential should agree to use an effective means of birth control.
10. Initial Required Laboratory Data:

    * ANC ≥ 1000/μL
    * Platelet count ≥ 100,000/μL
    * Serum Creatinine ≤ 2 mg/dL
    * Bilirubin ≤ 2 mg/dL
    * AST ≤ 2 x upper limit of normal

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2004-05; Primary Completion 2007-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Response | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Straus, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (47):
- United States (47):
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital at Howard Regional Health System, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - Iowa Blood and Cancer Care, Cedar Rapids, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Union Hospital Cancer Center at Union Hospital, Elkton MD, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - University of Minnesota Medical Center - Fairview, Minneapolis, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Saint Francis Cancer Treatment Center at Saint Francis Memorial Health Center, Grand Island, Nebraska
  - Great Plains Regional Medical Center, North Platte, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - CCOP - Hematology-Oncology Associates of Central New York, Syracuse, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Community General Hospital, Syracuse, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Lenoir Memorial Cancer Center, Kinston, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont

REFERENCES:
- [Result] Kostakoglu L, Straus DJ, Schöder H, et al.: Validation of the International Harmonization Project (IHP) Guidelines in early stage Hodgkin lymphoma (HL) treated with adriamycin, vinblastine and gemcitabine (AVG) (CALGB 50203): early results. [Abstract] Blood 112 (11): A-1460, 2008.
- [Result] Straus D, LaCase A, Juweid M, et al.: Doxorubicin, vinblastine and gemcitabine (AVG), a novel regimen excluding bleomycin for the treatment of early stage Hodgkin lymphoma (HL): results of CALGB 50203. [Abstract] Blood 110 (11): A-214, 2007.
- [Derived] Straus DJ, Johnson JL, LaCasce AS, Bartlett NL, Kostakoglu L, Hsi ED, Schoder H, Hall NC, Jung SH, Canellos GP, Schwartz LH, Takvorian RW, Juweid ME, Cheson BD; Cancer and Leukemia Group B. Doxorubicin, vinblastine, and gemcitabine (CALGB 50203) for stage I/II nonbulky Hodgkin lymphoma: pretreatment prognostic factors and interim PET. Blood. 2011 May 19;117(20):5314-20. doi: 10.1182/blood-2010-10-314260. Epub 2011 Feb 25. PMID 21355087